CLINICAL TRIAL: NCT03964025
Title: Clinical Investigation to Determine the Accuracy and Benefit of Cardioskin™ in Patients With Known Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: project stopped by the sponsor
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CL3-13001-002
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
Keywords: Holter Monitor; ECG Monitor; Cardioskin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardioskin™ and 3-lead Holter recorder (Experimental): This is single-arm study. All subjects will receive the investigational device (Cardioskin™) and comparator device (3-lead Holter recorder).The subject will be wearing both the Cardioskin™ and 3-lead Holter recorder for a period of 24 hours, after which the subject will continue wearing the Cardioskin™ alone for an additional period of 13 days.
  Interventions: Device: Wearing Cardioskin™ for 14 days

INTERVENTIONS:
Device: Wearing Cardioskin™ for 14 days — The current standard of care for diagnosing AF is through the use of a 24 hour Holter device. In this study, in addition to wearing the 3-lead Holter recorder for 24 hours, the subject will be wearing the Cardioskin™ for a period of 24 hours as well, after which the subject will continue wearing the Cardioskin™ alone for an additional period of 13 days.

SUMMARY:
This is a prospective, non-randomized, comparative, single-arm, open label, multi- centre, post-market clinical investigation involving an expected 74 subjects (minimum 40, maximum 118) suffering from paroxysmal AF with the aim to determine the accuracy of "definitive" AF detection (≥30 seconds) of the Cardioskin™ as compared to a 3-lead Holter recorder in patients with known paroxysmal AF.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, comparative, single-arm, open label, multi-centre, post-marketing clinical investigation involving an expected 74 subjects (minimum 40, maximum 118) suffering from paroxysmal AF. The clinical investigation will include a screening visit to determine subject eligibility, an inclusion visit where (additional) baseline characteristics will be collected and the subject will receive the investigational device (Cardioskin™) and comparator device (3-lead Holter recorder) (Visit 1), and 2 additional study visits. The subject will be wearing both the Cardioskin™ and 3-lead Holter recorder for a period of 24 hours, after which the subject will continue wearing the Cardioskin™ alone for an additional period of 13 days. The clinical investigation primarily aims to determine the accuracy of AF detection (≥30 seconds) of the Cardioskin™ wearable 15 lead ECG monitor as compared to a 3 lead Holter recorder in patients with known paroxysmal AF. Further objectives of the clinical investigation include detection of AF for the 13 additional days, detection of other arrhythmias and patient safety. A 3 lead Holter recorder was selected as the comparator device, because it is currently the gold standard for 24-hour home-based ECG monitoring.

ELIGIBILITY:
Inclusion Criteria:

The subject shall only be enrolled in the clinical investigation if he/she:

* is willing and able to understand and sign informed consent, and has signed an information and inform consent;
* is male or female;
* has a documented history of AF in the 3 months prior to screening e.g. by means of an ECG report, with at least one episode ≥30 seconds;
* has a subject reported frequency of at least one AF episode in the 48 hours prior to screening, as defined by AF related complaints;
* is on stable cardiovascular medication in the 2 weeks prior to screening and no changes to the cardiovascular medication are expected for the duration of the clinical investigation;
* has body weight characteristics that are compatible with the proposed models of Cardioskin™ (the subject fits the t-shirt);
* is minimum 18 years of age when signing informed consent;
* is willing and able to comply with the instructions outlined in the User Manual of the investigational device;
* is willing and able to comply with the instructions outlined in the User Manual of the Holter recorder (;
* is willing and able to comply to the schedule of assessment of the clinical investigation.

Exclusion Criteria:

The subject shall not be enrolled in the clinical investigation if he/she:

* has an implantable loop recorder; NOTE: this exclusion criterion is not applicable to all subjects in the clinical investigation. This exclusion criterion comes into effect once 4 subjects have been enrolled with an implantable loop recorder. This number of 4 may increase, to a maximum of 10% of enrolled subjects.
* has an implanted pacemaker or defibrillator;
* is lactating, pregnant, or planning to become pregnant during the course of the clinical investigation;
* is an alcohol and/or drugs abuser, on the investigator judgement and based on the patient questioning;
* has a known allergy to one of the components of the Cardioskin™ garment, including:

  * polyamide;
  * polyester;
  * elastane;
  * silicone;
  * silver;
  * any synthetic material.
* has a known allergy to ECG stickers;
* has a lot of chest hair;
* has a sensory disorder making the patient insensitive to pain on the skin;
* has behavioural problems making the patient excessively agitated or aggressive;
* has motor or mental disorders preventing the patient from expressing pain;
* has cardiorespiratory disorders which may be aggravated by the slight compression of the thorax;
* has an open wound on the skin, in the area either covered or surrounded by Cardioskin™ textile;
* has a strong contagious risk to any material composing Cardioskin™;
* is currently participating in, or has recently exited from (within 30 days prior to screening for this clinical investigation), or plans to be enrolled (during the course of this clinical investigation) in another clinical investigation.

In addition, subjects shall be excluded on sex (male/female) if an enrolment of 60% for one of the genders has been reached. At the end of the study, maximum 60% of the enrolled subjects shall be male and maximum 60% of the subjects shall be female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative likelihood ratio, positive and negative predicted value of recording "definite" AF episodes (≥30 seconds) with the Cardioskin™ versus 3-lead Holter recorder after a 24 hour recording period[performance]. | 24 hours
  Sensitivity, specificity, positive and negative likelihood ratio, and positive and negative predicted value of recording "definite" AF episodes (≥30 seconds) with the Cardioskin™ versus the 3-lead Holter recorder after a 24 hour recording period (adjudicated events)
The incidence of device related (serious) adverse events [safety]. | 14 days
  The incidence of device related (serious) adverse events during the course of the clinical investigation.

SECONDARY OUTCOMES:
Time until first "definite" AF (≥ 30 seconds) episode detection of the Cardioskin™. | 14 days
  Time until first "definite" AF episode detected by the Cardioskin™.
Incidence and length of AF episodes after 13 day recording period with Cardioskin™ (based on standard ECG analysis) | 13 days
  The incidence and length of AF episodes after a 13 day recording period, based on a standard ECG analysis, after first "definite" AF episode detected during this period.
Qualitative comparison of the relevant cardiac parameters as recorded by the Cardioskin™ to these recorded by a 3-lead holter, as assessed per standard ECG analysis after 24 hours. | 24 hours
  A qualitative comparison of the relevant cardiac parameters as recorded by the Cardioskin™ to these recorded by a 3-lead Holter recorder, assessed per standard ECG analysis.
The timing and frequency of subject reported AF episodes and timing, frequency and duration of AF episodes as detected by Cardioskin™ after 14 day recording period. | 14 days
  The timing and frequency of AF symptoms as recorded by the subject and the timing, frequency and duration of AF episodes as detected by the Cardioskin™ after a 14 day recording period.
Frequency and duration (total duration & longest) of arrhythmia symptoms as recorded by the subject and the nature, timing, frequency and duration (longest) of arrhythmia as detected by Cardioskin™ after a 14 day period(based on standard ECG analysis). | 14 days
  The timing and frequency of arrhythmia symptoms as recorded by the subject and the nature, timing, frequency and duration of arrhythmias as detected by the Cardioskin™ after a 14 day recording period, based on a standard ECG analysis.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Maastricht Universitair Medisch Centrum, Maastricht, Limburg
  - Universitair Medisch Centrum Groningen, Groningen
  - Martini Ziekenhuis, Groningen

IPD SHARING:
Plan to Share IPD: No